CLINICAL TRIAL: NCT07065747
Title: Objective Grading of Intraocular Inflammation in Uveitis Using Optical Coherence Tomography
Brief Title: Quantification & Classification of Inflammatory Cells in Uveitis Using OCT
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Professor, Oregon Health and Science University
Other Study IDs: OHSU IRB0008052; R21EY036563 (NIH)
Record Dates: First submitted 2025-07-02; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Anterior Uveitis (AU); Birdshot Chorioretinitis; Behcet Disease; Herpes Simplex Virus; Juvenile Idiopathic Arthritis (JIA); Spondyloarthritis (SA); Sarcoidosis; Posterior Vitreous Detachment
MeSH Terms: conditions — Uveitis, Anterior; Birdshot Chorioretinopathy; Behcet Syndrome; Herpes Simplex; Arthritis, Juvenile; Spondylarthritis; Sarcoidosis; Vitreous Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Uveitis Group: Eyes with active inflammation due to various systemic diseases
- Posterior Vitreous Detachment Group: Eyes with vitreous floaters and posterior vitreous detachment
- Healthy/Control Group: Healthy eyes with no history of uveitis, posterior vitreous detachment, or previous eye surgery

SUMMARY:
The goal of this study is to determine if it's possible to use a high resolution imaging device called optical coherence tomography (OCT) to develop an unbiased, standard method of counting and categorizing the various types of cells and proteins found in an eye condition called anterior uveitis. Anterior uveitis is a type of inflammation in the eye that can be caused by many different diseases of the body.

ELIGIBILITY:
Inclusion Criteria:

1. Uveitis Group: Eyes with active intraocular inflammation and a clinical diagnose of spondyloarthritis/HLA-B27 associated anterior uveitis, Juvenile Idiopathic Arthritis (JIA) associated chronic anterior uveitis, Herpes Simplex Virus (HSV) anterior uveitis, Birdshot chorioretinitis, Behcet disease uveitis, sarcoidosis associated uveitis, uveitis of any additional type, or uveitis masquerade.
2. Posterior Vitreous Detachment Group: Eyes with vitreous floaters and posterior vitreous detachment (PVD).
3. Healthy/Control Group: Healthy eyes with no history of uveitis, PVD, or previous eye surgery.

Exclusion Criteria:

1. Inability to give informed consent.
2. Inability to maintain stable fixation for OCT imaging.
3. Inability to commit to required visits to complete the study.
4. Pregnancy and breastfeeding.

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be recruited from clinical practices of the investigators at Casey Eye Institute of Oregon Health & Science University in Portland, Oregon.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Identification & Measurement of Anterior Chamber Cells | Day 1
  Anterior Chamber (AC) cells will be identified from OCT images by computer algorithms. AC cell number counted by OCT will be correlated with slit lamp grading. Cell size & other characteristics identified from OCT images will be associated with different uveitis diagnostic categories. The Standardization of Uveitis Nomenclature (SUN) grading system (scale: 0 = none to 4+ = severe) will be used to compare OCT-derived quantification against slit-lamp grading performed by attending physicians.

SECONDARY OUTCOMES:
Measure of AC Flare | Day 1
  OCT signal of the aqueous humor will be analyzed and correlated with slit lamp grading by the attending physician. The SUN grading system (scale: 0 to 4+) will be used.
Measure of Keratic Precipitates | Day 1
  Keratic precipitates (KPs) will be identified from OCT images. The size of the KPs will be compared across different uveitis diagnostic categories. There is no formal grading system for KPs. The investigators will use the typical qualitative assessments of morphology, distribution, and density. For morphology, cells will be described as fine, mutton-fat, stellate, or pigmented. Distribution patterns will be described as Arlt's Triangle, diffuse, central, or ring-shaped. Density will be described as few, moderate, or numerous.
Measure of Vitreous Cells | Day 1
  Vitreous cells will be identified from OCT images. Counting of vitreous cells will be done by computer algorithms. Since vitreous cells are not formally graded or quantified in the SUN system, physician grading will be described as rare, few, moderate, numerous, or sheets and compared against the OCT-derived measurements.
Measurement of Vitreous Haze | Day 1
  OCT signal of the vitreous clarity will be compared against clinical grading of vitreous haze. The National Eye Institute (NEI) Grading Scale will be used. Grading will be documented on a scale of 0 = no haze to 4+ = severe haze.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Casey Eye Institute - Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No